CLINICAL TRIAL: NCT02374268
Title: Intervention for Sarcopenia Among Older Chinese Adults: A Randomized Controlled Trial Assessing the Role of Exercise Program and Nutrition Supplement
Brief Title: Intervention Assessing the Role of Exercise Program and Nutrition Supplement for Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ruth Chan, Research assistant professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014.648-T
Record Dates: First submitted 2015-02-12; First posted 2015-02-27 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise program alone (Experimental): There will be 2 site sessions and 1 home session per week for 12 weeks. Each site exercise session will begin and end with a 5-10 minute warm-up and cool-down routine. The first part of the exercise program consists of 20-30 minute chair-based resistance exercises using Thera-Bands for muscle groups in both the upper and lower body. To target the development of muscle power in both the lower and upper extremities, participants will be instructed to perform each concentric movement 'as rapidly as possible,' and the eccentric movement in a slow and controlled manner. A 5-minute rest period will be given prior to the start of the second part of the exercise program that consists of aerobic exercises such as ball games using fitballs or Taichi. Participants will be asked to spend an hour/week on home exercise. Thera-Bands and a leaflet showing the exercise procedures will be given to them and their caregivers.
  Interventions: Behavioral: Exercise program alone
- Exercise program plus nutrition supplement (Experimental): This group will receive both the exercise program as well as the nutrition supplement. The components of the exercise program will be same as those of the exercise program alone group. Participants will also be asked to consume two sachets of Ensure NutriVigor every day during the 12-week intervention period. Ensure NutriVigor (one sachet of 54.1 g powder) contains 231 calories, 8.61 g protein, 1.21 g hydroxyl-methyl-butyrate (HMB), 130 IU vitamin D, and 0.29 g omega 3 fatty acid per serving. Participants will be instructed on how to prepare the supplement.
  Interventions: Behavioral: Exercise program alone; Dietary Supplement: Combined exercise program and nutrition supplement
- Waitlist control group (Other): This group will be asked to maintain their usual physical activities and dietary habits during the first 6 months of study period. After they complete the 24-week measurement, they will receive the same 12-week exercise program as of the exercise program alone group.
  Interventions: Other: Waitlist control group

INTERVENTIONS:
Behavioral: Exercise program alone
  Arms: Exercise program alone; Exercise program plus nutrition supplement
Dietary Supplement: Combined exercise program and nutrition supplement
  Arms: Exercise program plus nutrition supplement
Other: Waitlist control group
  Arms: Waitlist control group

SUMMARY:
Sarcopenia represents the loss of skeletal muscle and strength that occurs with aging. It is a major component of frailty and its effect on daily functioning, falls, and fractures has been well documented. Along with the population aging worldwide, the number of people with sarcopenia is expected to increase and, thus, contributing to dependency and the anticipated increase in health and social care costs. The cause of sarcopenia is multifactorial. Recent evidence suggests that some reversibility exists, highlighting the importance of intervention modalities. However, the role of nutritional supplementation and exercise programs, either individually or in combination, is still uncertain, and further randomized controlled trials (RCTs) have been recommended by the International Sarcopenia Initiative. Therefore, the investigators plan to conduct a 24-month RCT to compare the effectiveness of 12-week exercise program alone, combined exercise program and nutrition supplement, and non-exercise control group on improving muscle mass, strength and power and physical performance in Chinese older people who have sarcopenia defined using the Asian Working Group Criteria (AWGC). The investigators hypothesize that compared with the non-exercise control group, there will be improvement in muscle strength, power and mass, and physical performance in the exercise alone group, and that there will be an additive effect with the combined exercise and nutrition supplement group. Chinese older people aged 65 years and over will be recruited for a brief screening of sarcopenia and cognitive status. Potential subjects will further undertake detailed body composition and biochemical measurements to check for their eligibility. Eligible subjects will be randomized to one of the three groups: exercise program alone, combined exercise program and nutrition supplement, or waitlist control group with the same exercise program offered after 24-week of study enrollment. Each group will have 45 subjects. Outcome measurements including muscle strength, power and mass, physical performance, instrumental activities of daily living and related biochemical measurements will be made at baseline, 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chinese origin
* Normally reside in Hong Kong
* Could speak and understand Chinese
* With handgrip strength less than 26 kg for men and 18 kg for women and/or usual gait speed less than or equal to 0.8 m/s, as recommended by the Asian Working Group on Sarcopenia (AWGS)
* With height-adjusted appendicular skeletal muscle mass (ASM/ht2) measured using dual X-ray absorptiometry (DEXA) less than 7.0 kg/m2 for men and 5.4 kg/m2 for women, as recommended by the AWGS
* Willing to follow the study procedures

Exclusion Criteria:

* Recent (i.e. past 3 months) or concurrent participation in any clinical trial or dietary and/or exercise intervention program
* Self-reported allergy to the ingredients of the nutrition supplement
* Use of medications that could affect study outcomes
* With cancer conditions that are currently undergoing treatment
* Poorly controlled or unstable chronic obstructive pulmonary disease
* Poorly controlled or unstable cardiovascular disease or diabetes or hypertension
* Recent unhealed bone fracture (within the past 12 months)
* With medical advice or conditions prohibiting exercise or medical conditions that precluded safe participation in an exercise program
* With any other indication of a major medical or psychological illness, as judged by the investigators as ineligible to participate the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-03; Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Change in gait speed | baseline, 12 weeks
  This outcome will be measured using the 6-meter walk test

SECONDARY OUTCOMES:
Handgrip strength | baseline, 12 weeks
  Handgrip strength will be measured using a dynamometer
Bilateral leg extensors strength | baseline, 12 weeks
  Bilateral leg extensors strength will be measured by spring gauge while seated, and the average value between right and left will be used for analysis.
Muscle power in the upper extremities | baseline, 12 weeks
  This outcome will be measured using seated 1.8kg medicine ball throw test (maximum throw distance achieved in 3 trials).
Muscle power in the lower extremities | baseline, 12 weeks
  This outcome will be measured using 5-chair stand test (time to complete standing from a chair 5 times as quickly as possible).
Height-adjusted appendicular skeletal muscle mass | baseline, 12 weeks
  This outcome will be measured using dual X-ray absorptiometry (DEXA)
Improvement in sarcopenia category | baseline, 12 weeks
  This outcome will be measured using DEXA
Health-related quality of life | baseline, 12 weeks
  This outcome will be measured using validated Chinese version of short form (SF)-12
Instrumental Activities of Daily Living (IADL) | baseline, 12 weeks
  Participants will be asked to self-report of any impairment in walking two to three blocks outdoors on level ground, climbing 10 steps without resting, preparing own meals, doing heavy housework like scrubbing floors or washing windows, and shopping for groceries or clothes. A summed score from 0 to 5 was calculated from these activities as the degree of impairment in IADLs, with higher score indicating greater impairment.
Cardiorespiratory fitness | baseline, 12 weeks
  Cardiorespiratory fitness will be measured by 6-minute walk test (6MWT). 6MWT will be completed and scored as the total number of meters walked in 6 minutes.
Serum cystatin C measurement measured using immunoassay method | baseline, 12 weeks
  For combined exercise program and nutrition supplement group only
Renal function test measured by University Pathology Service | baseline, 12 weeks
  For combined exercise program and nutrition supplement group only

OTHER OUTCOMES:
Fasting blood samples for genetic study of genes related to physical function, sarcopenia and frailty | baseline, 12 weeks
Change in gait speed | 12 weeks, 24 weeks
  This outcome will be measured using the 6-meter walk test
Handgrip strength | 12 weeks, 24 weeks
  Handgrip strength will be measured using a dynamometer
Bilateral leg extensors strength | 12 weeks, 24 weeks
  Bilateral leg extensors strength will be measured by spring gauge while seated, and the average value between right and left will be used for analysis.
Muscle power in the upper extremities | 12 weeks, 24 weeks
  This outcome will be measured using seated 1.5kg medicine ball throw test (maximum throw distance achieved in 3 trials).
Muscle power in the lower extremities | 12 weeks, 24 weeks
  This outcome will be measured using 5-chair stand test (time to complete standing from a chair 5 times as quickly as possible).
Height-adjusted appendicular skeletal muscle mass | 12 weeks, 24 weeks
  This outcome will be measured using DEXA
Improvement in sarcopenia category | 12 weeks, 24 weeks
  This outcome will be measured using DEXA
Health-related quality of life | 12 weeks, 24 weeks
  This outcome will be measured using validated Chinese version of SF-12
Instrumental Activities of Daily Living | 12 weeks, 24 weeks
  Participants will be asked to self-report of any impairment in walking two to three blocks outdoors on level ground, climbing 10 steps without resting, preparing own meals, doing heavy housework like scrubbing floors or washing windows, and shopping for groceries or clothes. A summed score from 0 to 5 was calculated from these activities as the degree of impairment in IADLs, with higher score indicating greater impairment.
Cardiorespiratory fitness | 12 weeks, 24 weeks
  Cardiorespiratory fitness will be measured by 6-minute walk test (6MWT). 6MWT will be completed and scored as the total number of meters walked in 6 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Zhu LY, Chan R, Kwok T, Cheng KC, Ha A, Woo J. Effects of exercise and nutrition supplementation in community-dwelling older Chinese people with sarcopenia: a randomized controlled trial. Age Ageing. 2019 Mar 1;48(2):220-228. doi: 10.1093/ageing/afy179. PMID 30462162